CLINICAL TRIAL: NCT06531564
Title: Emergency Department Management of Isolated Femur Fracture Patients
Brief Title: Emergency Department Management of Femur Fractures
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: isolated femur fracture
Record Dates: First submitted 2024-07-17; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Femur Fracture; Pain, Joint; Analgesia
Keywords: isolated femur fracture; analgesia; emergency department; nerve block
MeSH Terms: conditions — Femoral Fractures; Arthralgia; Agnosia; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Opioid group: patients receiving intravenous opioid agents after femur fracture
- NSAID: patients receiving intravenous NSAID agents after femur fracture
- acetaminophen: patients receiving intravenous acetaminophen after femur fracture
- Femoral nerve block: patients receiving femoral nerve blocking treatment after femur fracture
- PENG block: patients receiving PENG blocking treatment after femur fracture

SUMMARY:
Comparison of emergency department management of patients presenting with isolated hip fracture: comparison of methods used in pain management, monitoring, and treatment; comparison of hospitalization durations; comparison of mortality

DETAILED DESCRIPTION:
Patient demographics, mechanism of injury, femur fracture classification, associated treatments, pre-procedural pain scoring, post-procedural pain scoring, orthopedic consultation, and patient outcomes (discharge, admission to ward or ICU, mortality) will be recorded on the data form.

For acute pain management, the timing of treatment administration, effectiveness of the applied method based on pre- and post-procedural pain scoring systems will be assessed. Post-procedural pain scores will be collected at 30, 60, and 120 minutes.

Long-term complications as a result of hospitalization following emergency department follow-ups will include monitoring on days 7 and 21 for mortality and morbidity.

The patients will be analyzed in 5 groups based on the treatments administered in the emergency department.

1. IV Opioid
2. IV NSAID
3. IV acetaminophen
4. Femoral nerve block
5. PENG block The researcher will not interfere with the treatment decision made by the responsible physician or the treatment process

ELIGIBILITY:
Inclusion Criteria:

Patients over the age of 18 years

Exclusion Criteria:

Forensic cases Patients who do not have follow-up in our healthcare system or cannot be followed up Patients with allergies to opioids or local anesthetics Patients with suspected neuropathy among defined complications of diabetes mellitus Patients requiring treatment for ≥2 different types of fractures upon emergency department admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients over the age of 18 years administered to emergency department with isolated femur fracture receving analgesia
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
effective analgesia after receiving treatment | 24 hours
  patients will be evaluated before and after analgesic treatments according to pain scales ( visual analogue scale, verbal pain intensity scale, PAINAD ( pain assessment in advanced dementia) scale andvisual analogue scale), effective pain management will be primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simic A, Nesek Adam V, Rosic D, Kocet N, Svetec M, Herceg A, Keranovic A, Rasic Z. PERIPHERAL NERVE BLOCKS FOR HIP FRACTURES IN EMERGENCY MEDICINE. Acta Clin Croat. 2022 Jun;61(Suppl 1):78-83. doi: 10.20471/acc.2022.61.s1.13. PMID 36304813
- [Background] Thiam CN, Khor HM, Pang GHM, Lim WC, Shanmugam T, Chandrasekaran CSK, Singh S, Zakaria MIB, Ong T. Hip fracture management in the emergency department and its impact on hospital outcomes: a retrospective cross-sectional analysis. Eur Geriatr Med. 2022 Oct;13(5):1081-1088. doi: 10.1007/s41999-022-00654-0. Epub 2022 May 14. PMID 35567676
- [Background] Fahey A, Cripps E, Ng A, Sweeny A, Snelling PJ. Pericapsular nerve group block for hip fracture is feasible, safe and effective in the emergency department: A prospective observational comparative cohort study. Emerg Med Australas. 2022 Dec;34(6):884-891. doi: 10.1111/1742-6723.14013. Epub 2022 Jun 14. PMID 35701386